CLINICAL TRIAL: NCT01550146
Title: Effects of a Single Dose of Dexamethasone in Patients Undergoing Operative Fixation of Proximal Femur Fracture
Brief Title: Single Dose of Dexamethasone in Femur Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cork University Hospital (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Principal Investigator, Szilard Szucs, Clinical Tutor in Anaesthesia, Cork University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14640820
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Fractured Neck of Femur
Keywords: Fractured neck of femur; Dexamethasone
MeSH Terms: conditions — Femoral Neck Fractures | interventions — dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone, 0.1 mg/kg (Experimental): The patients in the Dexamethasone group get iv 0.1 mg/kg dexamethasone preoperative.
  Interventions: Drug: Dexamethasone acetate
- Placebo (Placebo Comparator): In the Placebo group the patients get 0.1 ml/kg normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone acetate — iv. dexamethasone 0.1 mg/kg
  Arms: Dexamethasone, 0.1 mg/kg
Drug: Placebo — iv. Normal Saline 0.1 ml/kg
  Arms: Placebo

SUMMARY:
Fracture neck of femur is a common cause of hospital admission in the elderly and requires operative fixation.

Dexamethasone has the potential of inhibiting cortisol secretion. In addition, preoperative glucocorticoids improve analgesia and decrease opioid consumption with reduction in associated side effects in a variety of clinical settings.

The investigators hypothesis was that a single dose of preoperative dexamethasone enhance postoperative analgesia and attenuates the inflammatory response in patients undergoing operative fixation of fractured neck of femur, in a prospective, randomized, placebo controled trial.

DETAILED DESCRIPTION:
Having obtained ethical approval and written informed consent from each, 40 patients scheduled to undergo operative fixation of fractured neck of femur will be randomized using sealed envelopes to two groups.

Patients in the Dexamethasone group receive a single dose of 0.1 mg/kg dexamethasone iv. preoperative, patients in the Placebo group receive the same amount of Normal Saline. The anaesthetic technique is standardized, salive samples, blood samples are taken and pain scores are measured on a visual analog scale postoperatively at several timepoints.

ELIGIBILITY:
Inclusion Criteria:

* above 65 years
* ASA I-III patients

Exclusion Criteria:

* patient refusal
* outside age range
* coagulation disorders
* depression
* Cushing syndrome
* endocrine disorders
* corticosteroid treatment in the last 4 month
* head injury or associated injuries
* Mini Mental Scores < 25

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain scale at rest and on movement postoperatively | Postoperative in recovery, 6, 12, 24, 48, 72 hourly

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

REFERENCES:
- [Derived] Szucs S, Jessop D, Iohom G, Shorten GD. Postoperative analgesic effect, of preoperatively administered dexamethasone, after operative fixation of fractured neck of femur: randomised, double blinded controlled study. BMC Anesthesiol. 2016 Sep 22;16(1):79. doi: 10.1186/s12871-016-0247-5. PMID 27658581